CLINICAL TRIAL: NCT00812487
Title: Glycemic Control and Variability for Congestive Heart Failure Exacerbation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kathleen Dungan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Kathleen Dungan, Assistant Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008H0087; 1R21DK081877-01 (NIH)
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Results first posted 2013-12-31 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-11

CONDITIONS: Congestive Heart Failure; Diabetes Mellitus
Keywords: congestive heart failure; diabetes mellitus; hyperglycemia
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous insulin (Experimental)
  Interventions: Drug: Intravenous insulin
- Subcutaneous Insulin (Active Comparator): 4 injections of insulin/day
  Interventions: Drug: Subcutaneous insulin

INTERVENTIONS:
Drug: Intravenous insulin — Patients will receive continuous insulin infusion through the vein.
  Arms: Intravenous insulin
Drug: Subcutaneous insulin — 4 injections of insulin/day
  Arms: Subcutaneous Insulin

SUMMARY:
High glucose as well as fluctuations (rapid swings) in blood glucose can contribute to severe hospital complications and even death.

DETAILED DESCRIPTION:
High glucose as well as fluctuations in blood glucose can contribute to severe hospital complications and even death. Studies also suggest that heart failure patients who have high glucose or diabetes do not live as long as patients with normal glucose. Glucose fluctuations have not been well-studied in patients with heart failure. In this study, we will determine whether better control of blood sugar fluctuations in the hospital improve outcomes. We will enroll 80 patients with severe heart failure and divide them into 2 groups. We will use intravenous (given through the vein) insulin to lower blood sugar levels in group 1, and insulin injections (under the skin) in group 2. We will determine whether intravenous insulin improves blood markers of inflammation, changes in vital signs, and other tests that predict mortality in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Admitted (less than 48 hours) to the with worsening heart failure
* Hyperglycemia or diabetes. Hyperglycemia is defined as blood glucose greater than 150 mg/dL on at least 2 occasions separated by at least 4 hours apart, insulin use, or HbA1c >6.5%.

Exclusion Criteria:

* Type 1 diabetes
* Receiving comfort care measures only
* Hospital stay expected to be less than 2 days
* Pregnancy
* Prisoners
* Participation in the study on prior hospitalizations
* Acute myocardial infarction within 3 months
* End stage renal or liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-01; Primary Completion 2012-08 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Dungan, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospitalized patients with type 2 diabetes and heart failure exacerbation were recruited between 2008-2013 from an academic medical center.
Pre-assignment Details: Patients were randomized to intravenous or subcutaneous insulin. There were no pre-assignment changes in therapy before randomization. One patient was excluded after consent but prior to randomization due to receipt of corticosteroids which is an exclusion criterion.
Groups:
- Intravenous Insulin: Patients received intravenous insulin according to the hospital nursing run algorithm with a target glucose of 100-150 mg/dl.
- Subcutaneous Insulin: Patients received basal and bolus insulin, approximately 5 injections of insulin/day
Period: Overall Study
Arm/Group | Intravenous Insulin | Subcutaneous Insulin
Started | 32 | 42
Completed | 26 | 39
Not Completed | 6 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Transfer to ICU prior to intervention | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Patients were excluded from the analyses as described in "Participant Flow"
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Insulin | Subcutaneous Insulin | Total
Number analyzed (Participants) | 26 | 39 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 23 | 41
  >=65 years | 8 | 16 | 24
Age Continuous [Mean (Standard Deviation); unit: years] | 61 (9.6) | 61.3 (12.4) | 61 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 21
  Male | 18 | 26 | 44
Region of Enrollment [Number; unit: participants]
  United States | 26 | 39 | 65

OUTCOME MEASURES:

1. Secondary Outcome: High Frequency Heart Rate Variability
Description: High frequency heart rate variability (HF HRV)is a measure of cardiac autonomic tone. Electrocardiographic measures were obtained using a Bionex system (Mindware, Gahanna, OH). The electrocardiogram was performed in the standard lead II configuration. Software (Mindware, Gahanna, OH) was used to derive HF HRV. HF HRV was calculated using power spectral analysis.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: ms^2
Arm/Group | Intravenous Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 15 | 12
ms^2 | 15.5 [1.4 to 58] | 13.9 [2.7 to 207]

2. Secondary Outcome: Pre-ejection Period (PEP)
Description: Pre-ejection period (PEP) is the time between the onset of electrical depolarization of the ventricle and the opening of the aortic valve, a measure of sympathetic tone. It is obtained noninvasively using cardiac impedance obtained using a Bionex system (Mindware, Gahanna, OH). PEP is measured in milliseconds; lower values reflect higher sympathetic tone.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Intravenous Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 14 | 14
ms | 120 (24) | 117 (20)

3. Secondary Outcome: High Sensitivity C-reactive Protein (Hs-CRP)
Description: High sensitivity C-reactive Protein (hs-CRP) is a measure of inflammation. hsCRP (range 0-15 mg/L) was performed using Immunlite 1000 assay (Siemens; Erlangen, Germany).
Time Frame: 72 hours
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Intravenous Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 26 | 34
mg/dl | 10.5 [5.2 to 26] | 15.9 [8.3 to 32]

4. Secondary Outcome: Brain Natriuretic Peptide (BNP)
Description: Laboratory analyses were performed by the study institution's Clinical Research Center using standard commercial kits
Time Frame: 72 hours
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Intravenous Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 22 | 38
pg/ml | 360 [167 to 878] | 299 [135 to 713]

5. Secondary Outcome: Quality of Life
Description: Quality of Life was measured using the Minnesota Living with Heart Failure Questionnaire, which is a 21 question survey that uses a likert scale of 0-5. Each item asks over the past 4 weeks whether they have had a particular symptom of heart failure and to classify the response as no symptoms (0) to having the symptom very much (5). Responses are summed for a total score (0-105).
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intravenous Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 20 | 34
units on a scale | 50.5 [25 to 74.5] | 45 [22.5 to 71.5]

6. Secondary Outcome: Glycemic Lability Index (GLI)
Description: GLI is a measure of glycemic variability. GLI is the sum of the square of the difference between successive glucose measurements divided by the difference in time between measurements
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: (mg/dl)^2/hr*day-1
Arm/Group | Intravenous Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 24 | 34
(mg/dl)^2/hr*day-1 | 0.83 [0.31 to 1.44] | 0.66 [0.29 to 2.01]

7. Primary Outcome: Hospital Length of Stay
Description: Duration of hospitalization
Time Frame: participants were followed for the duration of hospital stay, median hospital stay 8 day
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Intravenous Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 26 | 39
days | 7 [5 to 10.5] | 8 [5 to 12]

8. Primary Outcome: Hospital Readmission
Description: All-cause hospital readmission within 30 days
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Intravenous Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 26 | 39
participants | 7 | 15

9. Secondary Outcome: Coefficient of Variation (CV)
Description: CV is a measure of glycemic variability
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: percentage (mean glucose/SD)
Arm/Group | Intravenous Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 24 | 33
percentage (mean glucose/SD) | 24.5 (10.2) | 18.6 (8.5)

10. Secondary Outcome: Mean Glucose
Description: mean sensor glucose
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Intravenous Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 24 | 33
mg/dl | 139 (23) | 169 (49)

ADVERSE EVENTS:
Arm/Group | Intravenous Insulin | Subcutaneous Insulin
Serious Adverse Events (participants affected / at risk) | 16/26 | 21/39
Other Adverse Events (participants affected / at risk) | 8/26 | 4/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Insulin (N=26) | Subcutaneous Insulin (N=39)
Death (Cardiac disorders) | 2 (2) | 2 (2) — 30 day death
Mechanical ventilation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) — Any mechanical ventilation during hospital stay
Infection (Infections and infestations) | 4 (4) | 6 (6) — Any new infection post-intervention
Arrhythmia (Cardiac disorders) | 2 (2) | 4 (4) — Any new arrhythmia (such as Ventricular tachycardia, atrial fibrillation) post-randomization
Acute Renal Failure (Renal and urinary disorders) | 6 (6) | 8 (8) — New hemodialysis or creatinine >2 mg/dl post-randomization
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Insulin (N=26) | Subcutaneous Insulin (N=39)
Hypoglycemia (Metabolism and nutrition disorders) | 8 (25) | 4 (11) — Hypoglycemia, defined as any capillary blood glucose <70 mg/dl during the intervention period (72 hours)

LIMITATIONS AND CAVEATS:
The study was limited by study drop-out. Sensor glucose values were reduced due to sensor failures, and cardiac assessments were limited due to a high number of patients with ectopy, arrhythmia or paced rhythms at baseline precluding analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No